CLINICAL TRIAL: NCT06848582
Title: A Single-Arm, Non-Blind Clinical Study on the Efficacy and Safety of Umbilical Cord Blood Natural Killer (NK) Cell Therapy for Children With High-Risk, Recurrent/Refractory Soft Tissue Sarcoma
Brief Title: Umbilical Cord Blood NK Cell Therapy for High-Risk Pediatric Soft Tissue Sarcoma: Efficacy and Safety Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Prof, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXEC-2025-001
Record Dates: First submitted 2025-02-07; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Soft Tissue Sarcoma (STS)
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NK Arm (Experimental): The treatment regimen involves 8 doses of NK cells injected at specific time points over 3 months, followed by a 3-year follow-up period.
  Interventions: Biological: umbilical cord blood NK cells

INTERVENTIONS:
Biological: umbilical cord blood NK cells — All subjects will receive Ex vivo Expanded and activated umbilical cord blood NK cells infusion.

SUMMARY:
This is a single-arm, open-label, non-blind, phase I/II clinical trial evaluating the safety and efficacy of umbilical cord blood natural killer (NK) cell in children with high-risk and relapsed/refractory soft tissue sarcoma (STS).

Objective:

Assess the safety and efficacy of NK cell in high-risk and relapsed/refractory STS patients.

Observe the pharmacokinetics and pharmacodynamics of NK cells in these patients.

Study Design:

Single-arm, open-label, non-blind design. 40 patients with high-risk and relapsed/refractory STS will receive the NK cell combined with other treatment .

The treatment regimen involves 8 doses of NK cells injected at specific time points over 3 months, followed by a 3-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, participants must meet all of the following criteria:

1. Give informed consent and sign a written informed consent form.
2. Age ≤ 18 years, no gender limitation.
3. Karnofsky (≥16 years) or Lansky (<16 years) (Appendix 2) performance status score of at least 50 (Appendix 2).
4. Diagnosis of high-risk and relapsed/refractory pediatric soft tissue sarcoma, confirmed by clinical criteria, and who have undergone prior comprehensive treatment (surgery, chemotherapy, radiation, and/or stem cell transplantation).
5. Estimated survival time of at least 12 weeks.
6. Complete recovery from all acute toxicities of prior anti-cancer chemotherapy, such as bone marrow suppression with recovery to grade I.
7. Myelosuppressive chemotherapy: at least 21 days after the last myelosuppressive chemotherapy (42 days if prior use of nitrosourea).
8. Experimental drugs or anti-cancer therapies other than chemotherapy: not used within 28 days prior to the planned start of NK cell immunotherapy. Must be fully recovered from the clinical significant toxicity of the therapy.
9. Hematopoietic growth factors: at least 14 days after the last administration of long-acting growth factor or 3 days after the last administration of short-acting growth factor.
10. X-ray therapy (XRT): at least 14 days after local palliative XRT (small field mouth) or at least 42 days after other substantive bone marrow (BM) irradiation, including prior radioactive iodine-131 meta-iodobenzylguanidine (131I-MIBG) treatment.
11. Stem cell transplantation without whole-body irradiation (TBI): no evidence of active graft versus host disease (GvHD), and at least 56 days after transplantation or stem cell transplantation.
12. Laboratory tests during the screening period must meet the following conditions:

    Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L (ANC ≥ 0.5 × 10^9/L if bone marrow involvement).

    Platelet count (PLT) ≥ 75 × 10^9/L (PLT ≥ 20 × 10^9/L if bone marrow involvement).

    Bilirubin ≤ 1.5 times the upper limit of normal (ULN). Creatinine ≤ 1.5 times the ULN (calculated according to the standard Cockcroft-Gault formula).

    ALT/AST ≤ 3 times the ULN (can be relaxed to 5 times the ULN if liver metastasis is present).
13. Ability to comply with outpatient treatment, laboratory monitoring, and necessary clinical visits during the study. For pediatric or adolescent participants, the parent/guardian must be able to understand, consent, and sign the study informed consent form (ICF) and applicable child consent form before initiating any protocol-related procedures. The participant will be able to express their consent (where applicable) under the consent of the parent/guardian.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for the study:

1. Presence of symptomatic brain metastasis (patients with brain metastasis treated and symptomatically stable for at least 2 months before enrollment are eligible, but must be confirmed to have no cerebral hemorrhage symptoms by cranial brain MRI, CT, or venous contrast).
2. History of or current cardiovascular disease, including ≥ II-grade myocardial ischemia or myocardial infarction, uncontrolled arrhythmia (including QTc interval ≥ 450 ms in men and ≥ 470 ms in women), or ≥ III-IV-grade heart failure according to the NYHA standard (Appendix 3) or left ventricular ejection fraction (LVEF) < 50% according to echocardiography.
3. History of or current interstitial lung disease.
4. Coagulation function abnormality (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or receiving anticoagulation or thrombolytic therapy.
5. Any venous or arterial thromboembolic event within 12 months prior to enrollment, including cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
6. Known hereditary or acquired bleeding and thrombotic tendency (e.g., hemophiliacs, coagulation dysfunction, thrombocytopenia, splenomegaly).
7. Long-term, untreated wounds or fractures (excluding pathologic fractures caused by tumor).
8. Major surgery or severe traumatic injury, fracture, or ulcer within 4 weeks prior to enrollment.
9. Factors that significantly affect the absorption of oral drugs, such as difficulty swallowing, chronic diarrhea, and intestinal obstruction.
10. History of abdominal fistula, gastrointestinal perforation, or peritonitis within the past 6 months.
11. Urinary routine showing ≥ ++ proteinuria, and confirmed 24-hour urine protein ≥ 1.0 g.
12. Presence of symptomatic serous cavity effusion requiring treatment (including pleural effusion, ascites, pericardial effusion); note: asymptomatic serous cavity effusion can be enrolled, symptomatic serous cavity effusion can be enrolled after active symptomatic treatment (not using anti-cancer drugs for serous cavity effusion treatment), and eligible for enrollment according to the judgment of the researcher.
13. Active infection requiring anti-microbial therapy (e.g., requiring the use of antibacterial drugs, antiviral drugs, but not including chronic hepatitis B anti-hepatitis B treatment, anti-fungal drug treatment).
14. History of substance abuse of psychiatric drugs and inability to quit or with psychiatric disorders.
15. Participation in other anti-tumor drug clinical trials within the past 4 weeks.
16. Receiving systemic hormone treatment or other forms of immunosuppressive treatment within 2 weeks prior to the first dose of the study drug.
17. History of active autoimmune disease requiring systemic treatment (e.g., using disease-modifying drugs, corticosteroids, or immunosuppressive agents) within the past 2 years; note: alternative treatment (e.g., thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction) is not considered systemic treatment.
18. Contraindications for IL-2 use.
19. Active infection requiring systemic venous treatment.
20. Administration of live vaccines within 1 month prior to the first use of the study drug; live vaccines against seasonal influenza, injectable inactivated virus vaccines are allowed, but nasal administration of live attenuated influenza vaccines is not allowed.
21. Prior or concurrent other untreated malignant tumors, excluding cured superficial basal cell carcinoma, cervical in situ carcinoma, and superficial bladder carcinoma.
22. Other conditions judged by the researcher to potentially affect the conduct of the clinical research and the determination of research results.
23. Viral screening during the screening period showing any of the following:

    HBsAg positive and HBV DNA above the normal upper limit. Anti-HCV positive and HCV RNA positive. HIV positive.
24. Prior allogeneic tissue/organe transplantation.
25. Poor compliance, unable to cooperate with clinical research.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | Two weeks after the second cycle (a total of 16 weeks after the strart of first umbilical cord blood natural killer cell infusion)
  ORR was evaluated according to the International Neuroblastoma Response Criteria (INRC)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Dongguan Taixin Hospital, Dongguan